CLINICAL TRIAL: NCT03642288
Title: The Use of Gastrografin in Chronic Radiation Enteropathy With Small Bowel Obstruction：A Retrospective Study
Brief Title: The Use of Gastrografin in Chronic Radiation Enteropathy With Small Bowel Obstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Ding Chao, Clinical Doctor, Jinling Hospital, China
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Gastrografin-CRE
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: CRE-induced SBO
MeSH Terms: interventions — Diatrizoate Meglumine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRE-induced SBO (Experimental): Patients with CRE-induced SBO received GG challenge.
  Interventions: Drug: Gastrografin
- ASBO (Active Comparator): Patients with adhesive SBO (ASBO) received GG challenge.
  Interventions: Drug: Gastrografin

INTERVENTIONS:
Drug: Gastrografin — Patients with CRE-induced SBO or ASBO both received GG challenge.

SUMMARY:
Chronic radiation enteropathy (CRE) is a major issue for long-term cancer survivors. The aim of this study was to clarify the diagnostic and therapeutic effect of the Gastrografin (GG) challenge for patients with CRE induced small bowel obstruction SBO.

ELIGIBILITY:
Inclusion Criteria:

* with a first diagnosis of CRE combined with SBO and ASBO that was determined by clinical history, computed tomography (CT) manifestation, and conﬁrmed by intraoperative and histologic ﬁndings.
* radiation therapy completed at least 6 months before enrolment.

Exclusion Criteria:

* a colostomy or ileostomy;
* large bowel obstruction;
* with a known history of either allergy or hypersensitivity to iodinated contrast agents;
* with signs of strangulation;
* metastatic disease;
* obstruction within 4 weeks after a recent operation or serious comorbidity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
The rate of successful conservative treatment | 5 days
  The rate of patients who need for operative intervention within 48 hours of randomization.

SECONDARY OUTCOMES:
The time to resolution | 2 weeks
  The time to resolution of ASIO (flatus and bowel motion).
The length of hospital stays | 2 weeks
  The length of hospital stays (in hours, calculated from the hospital admission to resolution of intestinal obstruction).